CLINICAL TRIAL: NCT04521140
Title: Assessing eFficacy and Safety of DEXTENZA 0.4 mg inseRt in Conjunction With Topical Prednisolone Acetate 1% Treating Pain, and inflamMation Following Corneal Transplant Surgery Compared to Topical Prednisolone Acetate 1%.
Brief Title: Assessing eFficacy and Safety of DEXTENZA 0.4 mg inseRt, Following Corneal Transplant Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nicole Fram M.D. (Other)
Responsible Party: Sponsor-Investigator, Nicole Fram M.D., Principal Investigator, Advanced Vision Care
Organization: Advanced Vision Care (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVC-002
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Corneal Edema; Corneal Defect; Corneal Transplant; Penetrating KeratoPlasty; Anterior Chamber Inflammation; Ocular Pain; Intraocular Pressure
MeSH Terms: conditions — Corneal Edema; Eye Pain | interventions — Calcium Dobesilate; prednisolone acetate; Methylprednisolone

STUDY DESIGN:
Intervention Model Description: In patient who undergo corneal transplant (PKP,DSEK,DMEK), subjects will be randomized to 6 arms and be followed for a period of 3 months.
  First arm will Receive Dextenza with PKP, Second arm will receive Prednisolone Acetate 1% with PKP, Third arm will Receive Dextenza with DSEK, Forth arm will receive Prednisolone Acetate 1% with DSEK Fifth arm will Receive Dextenza with DMEK, Sixth arm will receive Prednisolone Acetate 1% with DMEK
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- PKP with Dextenza (study) (Experimental): Patients undergoing PKP will receive Dextenza insert with:
  topical prednisolone acetate 1% 4 times a day for 1 month, 3 times a day for one month, 2 times a day for one month, once a day for one month, then Lotemax once a day thereafter.
  PolymyxinB/Trimethoprim or Vigamox / Moxifloxacin 4 times a day for 2 weeks
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert; Drug: Prednisolone Acetate 1% Oph Susp
- PKP without Dextenza (Controlled) (Other): Patients undergoing PKP will receive:
  topical prednisolone acetate 1% every two hours (6X /day) for 2 weeks, 4 times a day for 1 month, 3 times a day for one month, 2 times a day for one month, once a day for one month, then Lotemax once a day thereafter.
  PolymyxinB/Trimethoprim or Vigamox / Moxifloxacin 4 times a day for 2 weeks
  Interventions: Drug: Prednisolone Acetate 1% Oph Susp
- DSEK with Dextenza (study) (Experimental): Patients undergoing DSEK will receive Dextenza insert with:
  topical prednisolone acetate 1% 4 times a day for 1 month, 3 times a day for one month, 2 times a day for one month, once a day for one month, then Lotemax once a day thereafter.
  PolymyxinB/Trimethoprim or Vigamox / Moxifloxacin 4 times a day for 2 weeks
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert; Drug: Prednisolone Acetate 1% Oph Susp
- DSEK without Dextenza (Controlled) (Other): Patients undergoing DSEK will receive:
  topical prednisolone acetate 1% every two hours (6X /day) for 2 weeks, 4 times a day for 1 month, 3 times a day for one month, 2 times a day for one month, once a day for one month, then Lotemax once a day thereafter.
  PolymyxinB/Trimethoprim or Vigamox / Moxifloxacin 4 times a day for 2 weeks
  Interventions: Drug: Prednisolone Acetate 1% Oph Susp
- DMEK with Dextenza (study) (Experimental): will receive Dextenza insert with: topical prednisolone acetate 1% 4 times a day for 1 month, 3 times a day for one month, 2 times a day for one month, once a day for one month, then Lotemax once a day thereafter.
  PolymyxinB/Trimethoprim or Vigamox / Moxifloxacin 4 times a day for 2 weeks
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert; Drug: Prednisolone Acetate 1% Oph Susp
- DMEK without Dextenza (Controlled) (Other): Patients undergoing DMEK will receive:
  topical prednisolone acetate 1% every two hours (6X /day) for 2 weeks, 4 times a day for 1 month, 3 times a day for one month, 2 times a day for one month, once a day for one month, then Lotemax once a day thereafter.
  PolymyxinB/Trimethoprim or Vigamox / Moxifloxacin 4 times a day for 2 weeks
  Interventions: Drug: Prednisolone Acetate 1% Oph Susp

INTERVENTIONS:
Drug: Dextenza 0.4Mg Ophthalmic Insert — DEXTENZA is a corticosteroid intracanalicular insert placed in the punctum, a natural opening in the eye lid, and into the canaliculus and is designed to deliver dexamethasone to the ocular surface for up to 30 days without preservatives.
  Other Names: Dexamethasone Ophthalmic Insert
  Arms: DMEK with Dextenza (study); DSEK with Dextenza (study); PKP with Dextenza (study)
Drug: Prednisolone Acetate 1% Oph Susp — Prednisolone Acetate 1% is a corticosteroid used as a topical drop after corneal transplant to decrease inflammation and prevent graft rejection
  Other Names: Omnipred, Pred Forte

SUMMARY:
Assessing the efficacy and safety of DEXTENZA, sustained release dexamethasone 0.4 mg insert following corneal transplant surgery (PKP, DSEK, DMEK) as compared to topical prednisolone acetate 1%.

DETAILED DESCRIPTION:
Assessing the efficacy and safety of DEXTENZA, sustained release dexamethasone 0.4 mg insert, when placed within the lower or upper eye lid canaliculus in conjunction with topical prednisolone acetate 1% for the treatment of pain, and inflammation following corneal transplant surgery (PKP, DSEK, DMEK) as compared to topical prednisolone acetate 1%.

ELIGIBILITY:
Inclusion Criteria: A patient's study eye must meet the following criteria to be eligible for inclusion in the study:

* Age 18 years and older
* Scheduled corneal transplant surgery: PKP, DSEK, DMEK
* Willing and able to comply with clinic visits and study related procedures
* Willing and able to sign the informed consent form

Exclusion Criteria: A patient who meets any of the following criteria will be excluded from the study:

* Patients under the age of 18.
* Pregnancy (must be ruled out in women of child-bearing age with pregnancy test)
* Active infectious systemic disease
* Active infectious ocular or extraocular disease
* Presence of punctal plug in the study eye
* Obstructed nasolacrimal duct in the study eye(s)
* Hypersensitivity to dexamethasone or prednisolone eye drops
* Patients being treated with immunomodulating agents in the study eye(s)
* Patients being treated with immunosuppressants and/or oral steroids
* Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Mean change in pain score | Assessed on Day 1,7 and 30
  as measured with the visual analog scale (VAS); between 0 and 100; 0 meaning no pain and 100 meaning worst pain possible
Mean change in inflammation (Cell and Flare) scores | Assessed on Day 1,7 and 30
  as measured by SUN (Standardization on Uveitis Nomenclature) grading scale: absence of cell to be defined as a grade of 0-0.5 and absence of flare to be defined as a grade of: 0-1

SECONDARY OUTCOMES:
Mean change in duration to corneal re-epithelization | Assessed on Day 1 and 7
  as measured by clinical observation of percentage (%); between 0 to 100%; 0 meaning complete re-epithalization and 100% meaning total corneal defect
Mean change in size of epithelial defect | Assessed on Day 1 and 7
  as measured by diameter (mm) of defect; 0 meaning no defect
Impact on the practice/medical team of decreasing the drop burden | Assessed on day 30
  as measured by a questionnaire
Mean change in duration to clearing of corneal edema | Assessed on Day 30, 60 and 90
  as measured by clinical observation; between 0 to 3; 0 meaning clear cornea and 3+ meaning complete obscuration of anterior chamber and iris

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Fram, MD, Principal Investigator — Advanced Vision Care
Locations (1):
- Advanced Vision Care, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anshu A, Price MO, Price FW Jr. Risk of corneal transplant rejection significantly reduced with Descemet's membrane endothelial keratoplasty. Ophthalmology. 2012 Mar;119(3):536-40. doi: 10.1016/j.ophtha.2011.09.019. Epub 2012 Jan 3. PMID 22218143
- [Background] Price MO, Scanameo A, Feng MT, Price FW Jr. Descemet's Membrane Endothelial Keratoplasty: Risk of Immunologic Rejection Episodes after Discontinuing Topical Corticosteroids. Ophthalmology. 2016 Jun;123(6):1232-6. doi: 10.1016/j.ophtha.2016.02.001. Epub 2016 Mar 13. PMID 26983976
- [Background] Tyson SL, Bafna S, Gira JP, Goldberg DF, Jones JJ, Jones MP, Kim JK, Martel JM, Nordlund ML, Piovanetti-Perez IK, Singh IP, Metzinger JL, Mulani D, Sane S, Talamo JH, Goldstein MH; Dextenza Study Group. Multicenter randomized phase 3 study of a sustained-release intracanalicular dexamethasone insert for treatment of ocular inflammation and pain after cataract surgery. J Cataract Refract Surg. 2019 Feb;45(2):204-212. doi: 10.1016/j.jcrs.2018.09.023. Epub 2018 Oct 24. PMID 30367938